CLINICAL TRIAL: NCT05590507
Title: A Remote Mindfulness-Based Physical Activity Intervention for Postmenopausal Women
Brief Title: Remote Mindfulness-Based Physical Activity Intervention for Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Emma Fortune Ngufor, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-007713
Record Dates: First submitted 2022-10-19; First posted 2022-10-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Postmenopausal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A/Intervention (Experimental): Subjects will use mindfulness audio recordings along with their physical activity, and will receive a weekly health coaching phone call along with supplemental educational materials.
  Interventions: Behavioral: Mindfulness Audio Recordings
- Group B/Control (No Intervention): Subjects will receive education materials on healthy habits for increasing physical activity based on the National Institutes of Health, and bi-weekly check-in phone call.

INTERVENTIONS:
Behavioral: Mindfulness Audio Recordings — A 5-minute audio file aimed to increase likelihood of experiencing positive affect associated with physical activity. Participants will listen to a mindfulness audio file at the beginning of each physical activity session they choose to engage in during weeks 2-4
  Arms: Group A/Intervention

SUMMARY:
The purpose of this study is to figure out if postmenopausal women find a mindfulness audio recording acceptable for use along with physical activity, and to find out if this tool is helpful in increasing daily physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients self-report as being > 1 year postmenopausal.
* Patients are able to walk without a walking aid.
* Patients own and know how to operate a smart phone or tablet.
* Patients are willing and able to complete the activity monitoring.
* Patients are self-reportedly underactive.

Exclusion Criteria:

* Patients are < 1 year postmenopausal.
* Patients require a walking aid for daily mobility.
* Patients do not own a smartphone or table, or are unwilling to use such a device for the purposes of the study.
* Patients' primary form of exercise is swimming (the activity monitors are not waterproof).
* Patients are unable or unwilling to complete activity monitoring.
* Patients are unable to provide informed consent independently.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Acceptability of a mindfulness-based physical activity intervention | 4 weeks
  Number of subjects to rate the remotely-accessible and physical activity-targeted mindfulness audio file as acceptable

SECONDARY OUTCOMES:
Daily physical activity | 4 weeks
  Number of subjects to have an increase in objectively measured daily physical activity variables (such as step counts) recorded by ActiGraph activity monitor

CONTACTS AND LOCATIONS:
Overall Officials: Emma Fortune-Ngufor, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No